CLINICAL TRIAL: NCT04086654
Title: Psychometric Properties of the International Trauma Interview (ITI) for ICD-11 PTSD and CPTSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ITI Project
Record Dates: First submitted 2019-09-09; First posted 2019-09-11 (Actual); Last update posted 2022-11-22 (Actual); Status verified 2022-11

CONDITIONS: Post Traumatic Stress Disorder (PTSD); Complex Post-Traumatic Stress Disorder (CPTSD)
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- International Trauma Interview (ITI) (Other)
  Interventions: Diagnostic Test: International Trauma Interview (ITI) for ICD-11 PTSD and Complex PTSD - German version

INTERVENTIONS:
Diagnostic Test: International Trauma Interview (ITI) for ICD-11 PTSD and Complex PTSD - German version — The ITI consists of 18 items and for each symptom, standardized questions as well as probes are presented. A trained professional rates both symptom frequency and intensity, which are converted into an overall index of symptom severity. A diagnosis of PTSD/CPTSD is established by applying the ICD-11 diagnostic rules. It takes approximately 30-60 minutes to administer.

SUMMARY:
The aim of the project is to evaluate the psychometric properties (e.g. validity, reliability) of the International Trauma Interview (ITI) - German version. The ITI is a structured clinical interview that corresponds to the ICD-11 criteria for diagnosing both posttraumatic stress disorder (PTSD) and complex posttraumatic stress disorder (CPTSD).

Eligible participants from psychiatric inpatient and outpatient facilities in Switzerland who have provided informed will complete various self-report measures about trauma-related mental health complaints. In addition, the ITI will be conducted by a trained clinician. Lastly, information from the medical chart will be further used for scientific purpose. The overall assessment will take approximately 1-2 hours to complete.

ELIGIBILITY:
Study-specific Inclusion criteria

* Structured diagnostic procedures upon hospital entry not yet started, except for orienting assessments
* Able to give informed consent as documented by signature
* Able to understand and communicate in German Exclusion criteria
* Clinical signs for impaired cognitive abilities
* Other contraindications to undergo the clinical interview

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2020-03-02 (Actual); Primary Completion 2021-10-15 (Actual); Study Completion 2021-10-15 (Actual)

PRIMARY OUTCOMES:
International Trauma Interview (ITI) | Up to two weeks upon psychiatric ward entry
Life Event Checklist DSM-5 | Up to two weeks upon psychiatric ward entry

SECONDARY OUTCOMES:
Beck Depression Inventory II | Up to seven days upon psychiatric ward entry
Brief Symptom Checklist | Up to seven days upon psychiatric ward entry
Impact of Event Scale Revised Version | Up to seven days upon psychiatric ward entry
PTSD Checklist for DSM-5 | Up to seven days upon psychiatric ward entry
Borderline Symptom List | Up to seven days upon psychiatric ward entry

CONTACTS AND LOCATIONS:
Locations (1):
- Integrierte Psychiatrie Winterthur, Spezialstation für Traumafolgestörungen, Winterthur, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Information about ICD-11 PTSD/CPTSD measures — https://www.traumameasuresglobal.com/itq
- See also: Chair organizing the study — https://www.psychology.uzh.ch/en/areas/hea/psypath.html